CLINICAL TRIAL: NCT06556758
Title: Effects of Stripping Massage on Rhomboid Major and Minor Active Trigger Points in Patients With Upper Thoracic Pain.
Brief Title: Stripping Massage on Rhomboid Major and Minor Active Trigger Points in Upper Thoracic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aqsa Mustafa
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Upper Thoracic Pain Due to Active Trigger Points
Keywords: Stripping massage, Upper thoracic pain, Active trigger points
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stripping massage + conventional Therapy (Experimental): Stripping Massage Stripping massage on rhomboid major and minor active trigger point in the direction of muscle fiber from origin to insertion of muscle. Frequency: 3 minutes for 3 times/week for 4 consecutive weeks.
  Conventional therapy including Hot pack for 10 minutes + ischemic compression for 90 secs + CPA glides grade 3 kaltenborn mobilization on thoracic T1 to T4 (5 reps x 1 set) Frequency: 3 times/ week for 4 weeks
  Interventions: Other: stripping massage + conventional therapy
- Conventional therapy (Active Comparator): Conventional Therapy Conventional PT including Hot pack for 10 minutes + ischemic compression for 90 secs + CPA glides grade 3 kaltenborn mobilization on thoracic T1 to T4(5 reps x 1 set ) Frequency : 3 times/ week for 4 weeks
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: stripping massage + conventional therapy — Stripping massage on rhomboid major and minor active trigger point in the direction of muscle fiber from origin to insertion of muscle. Frequency: 3 minutes for 3 times/week for 4 consecutive weeks. Conventional PT including Hot pack for 10 minutes + ischemic compression for 90 secs + CPA glides grade 3 kaltenborn mobilization on thoracic T1 to T4 (5 reps x 1 set) Frequency: 3 times/ week for 4 weeks
  Other Names: Stripping massage on rhomboid major and minor active trigger points
  Arms: stripping massage + conventional Therapy
Other: Conventional therapy — conventional therapy including Hot pack for 10 minutes + ischemic compression for 90 secs + CPA glides grade 3 kaltenborn mobilization on thoracic T1 to T4 (5 reps x 1 set ) Frequency : 3 times/ week for 4 weeks
  Arms: Conventional therapy

SUMMARY:
Aim of this randomized controlled trial is to see the effects of stripping massage on rhomboids major and minor active trigger points in patients with upper thoracic pain for reducing pain, enhancing thoracic range of motion and physical functioning

DETAILED DESCRIPTION:
Spine pain is a common condition that results in considerable levels of disability and lost work time and has a major impact on society, a lifetime prevalence ranging from 15.6% to 19.5% for thoracic pain. Thoracic pain is more prevalent in women than in men (2:1). The origin of spine pain is clearly multifactorial and often includes number of anatomical structures. One plausible etiology of symptoms associated with thoracic pain may be the presence of myofascial pain. Myofascial pain is generally associated with the presence of trigger points. Trigger points are hypersensitive spots within taut bands of skeletal musculature whose stimulation can be associated with referred pain and autonomic phenomena. Trigger points can be either active or latent depending on the association with symptoms. For instance, active trigger points (MTrPs) are associated with spontaneous pain, and the local and referred pain reproduces the symptoms of the patient, totally or partially.

Stripping massage (SM) is a gliding tissue massage technique that focuses on the deeper layers of the fascia and skeletal muscle.This technique involves gliding pressure along a muscle, usually from one attachment to the other in the direction of the muscle fibers. Applying SM to tender spots in muscles can cause ischaemia followed by reflexive hyperaemia. This increases the local blood flow, which improves pliability of the muscles and fascia and helps break down adhesions and decrease pain sensations. SM acts as a mechanical stress that stimulates parasympathetic activity which leads to the release of substances such as endorphins. These chemicals remove the noxious stimulus and decrease the pressure on nociceptors, reducing pain The rationale for the use of this technique is to identify the effects of stripping massage on rhomboids active trigger points in upper thoracic pain patients. This study will see the effects of stripping massage on rhomboids trigger points on pain, thoracic mobility, and functional performance. Aim of this study is to see the effects of stripping massage to figure out whether this technique would be more effective and should be incorporated into clinical settings in relation to conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.

  * females
  * Age: 18-40
  * Active TrPs in the rhomboid major and minor muscles.
  * Presence of atleast one trigger point in rhomboids (diagnosed by the characteristics like hyperirritable spot in a taut band, twitch response and referral pain)
  * Presence of Jump sign
  * Segmental hypomobility in upper thoracic region identified with positive springing test
  * upper thoracic pain, defined as pain in the body region encompassing from T1 to T4) pain intensity score of ≥ 3 on the numeric pain rating scale (0-10)
  * symptoms provoked by thoracic movement,or palpation of the rhomboid muscles.

Exclusion Criteria:

* Participants falling in this category would be excluded from the study.

  * a history of neck trauma
  * previously had surgery in the neck or shoulder area or suffered from physical injury
  * Fractures, Dislocations, Traumatic injuries, Adhesive capsulitis, thoracic outlet syndrome.
  * any rheumatic condition, osteoporosis, cancer, spinal infection, radicular pain, or neuropathy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale NPRS | 4 weeks
  The NPRS is a segmented numeric version of the visual analog scale which is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.

SECONDARY OUTCOMES:
Bubble inclinometer | 4 weeks
  It is an instrument that measures the available range of motion at a joint.

OTHER OUTCOMES:
Functional rating index | 4 weeks
  The Functional Rating Index (FRI) is an instrument specifically designed to quantitatively measure the subjective perception of function and pain of the spinal musculoskeletal system in a clinical environment

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Ali, MSOMPT, Principal Investigator — Riphah International University; Aqsa Mustafa, MSompt*, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No